CLINICAL TRIAL: NCT05643313
Title: Clinical Investigation on Feasibility and Usability of the ABLE Exoskeleton Device for Individuals With Spinal Cord Injury to Perform Skills for Home and Community Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: University Hospital Heidelberg (Other); Institut Guttmann (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABLEexoSCI Home
Record Dates: First submitted 2022-11-25; First posted 2022-12-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Exoskeleton; Robotics; Gait Rehabilitation; Lower-limb; Neurorehabilitation; Paraplegia; Walking; Assistive technology; Usability; Feasibility; Home use; Community use; Multicenter
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will then undergo a training programme with the ABLE Exoskeleton three to five times a week for up to 8 weeks for a total of 18 training sessions and 4 assessment sessions.
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — The ABLE Exoskeleton is a lower-limb overground robotic exoskeleton intended for SCI patients for rehabilitation in a clinical setting.

SUMMARY:
The loss of the ability to walk and the associated restriction of mobility presents a major challenge to people with spinal cord injury in an everyday environment designed for pedestrians. Exoskeletal technology has the potential to help people with impaired leg function to regain ambulation and thus improve their independence. This technology is not completely new, but due to their high access price (~120k€/unit), high size and weight (~25 kg), and need for trained physiotherapist supervision, commercially available exoskeletons are only found in large hospitals and only in very few cases get into patients' homes.

The company ABLE Human Motion S.L. (Barcelona, Spain) has developed a novel exoskeleton to overcome these disadvantages, which is more compact, lighter and easier to use.

The primary objective of this study is to determine the feasibility and usability of the ABLE Exoskeleton for persons with SCI to perform skills in home and community environments.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the feasibility and usability of the ABLE Exoskeleton for persons with SCI to perform skills for home and community environments during a training programme of up to 8 weeks. Results will be used to assess the potential of the device to be used in a home and community setting by persons with SCI, while providing meaningful insights to develop future features to improve its performance in those environments.

The secondary objectives are as follows:

* Assess the impact of ABLE Exoskeleton training on gait and function.
* Assess the effect of the ABLE Exoskeleton on the patients' perceived rate of exertion.
* Assess the impact of the ABLE Exoskeleton on the quality of life and general health of the participants.
* Assess the level of user satisfaction from participants and therapists of the ABLE Exoskeleton.
* Assess the psychosocial impact of the ABLE Exoskeleton for participants.

The primary hypothesis of this study is that the ABLE Exoskeleton is feasible to be used by persons with SCI to perform skills for home and community environments.

The secondary hypothesis is that the device will have a positive impact on the perceived rate of exertion, mobility and psychosocial health, and quality of life and general health of the study participants with SCI.

This is a multicenter pre-post quasi-experimental study. The pre-post period will cover 22 exoskeleton sessions (18 training sessions and 4 assessment sessions) over a period of up to 8 weeks. The study will have two centres specialized in SCI involved, one at Heidelberg University, Germany and another at Institut Guttmann, Spain. In total 10 patients will be recruited.

After obtaining a Patient Information Sheet and Informed Consent Form (PIS/ICF), patients will be screened. Patients who match inclusion and exclusion criteria and pass pre-study screening, will be enrolled into the study. First, there will be a familiarisation session (session 0), where participants will learn how to use the device. Participants will then undergo a training programme with the ABLE Exoskeleton three to five times a week for up to 8 weeks for a total of 18 training sessions and 4 assessment sessions. The assessment sessions with the device will be performed at 4 time-points throughout training: Baseline (Session 1), Mid-training (Session 11), Final-training (Session 21) and Home-Skills-Test (Session 22). This therefore means there will be a total of 22 exoskeleton sessions, including training and assessments. During each training session, feasibility measurements will be taken via the evaluation of the performance of exoskeleton skills. Four weeks after the post-training assessment, a follow-up assessment will be conducted with participants. At the end of the study, the participating therapists will be asked to fill out a satisfaction questionnaire.

ELIGIBILITY:
Participants will be taken from former or current patients at one of the two SCI centres.

Inclusion Criteria:

* 18 to 70 years of age
* Traumatic and non-traumatic SCI
* Motor incomplete SCI with Neurological Level of Injury (NLI) C5-L5, or, Motor Complete SCI with NLI T1-L5
* Time since onset of SCI > 6 months
* Ability to give informed consent

Exclusion Criteria:

* WISCI II without exoskeleton of >13
* 5 or more risk factors present for fragility as stated by Craven et al (Craven et al., 2009a).
* History of lower limb fragility fractures in the last 2 years
* Deterioration > 3 points of the total ISNCSCI motor score within the last 4 weeks
* Spinal instability
* Modified Ashworth scale 4 in lower limbs
* Unable to tolerate 30 min standing without clinical symptoms of orthostatic hypotension
* Unable to perform a sit-to-stand transfer or stand in the device with assistance
* Psychological or cognitive issues that do not allow the participant to follow the study procedures
* Known pregnancy or breastfeeding
* Any neurological condition other than SCI
* Medically unstable - Unstable cardiovascular system, hemodynamic instability, untreated hypertension (Systolic blood pressure > 140, Diastolic blood pressure > 90 mmHg), unresolved DVT, uncontrolled autonomic dysreflexia.
* Severe comorbidities - Any condition that a physician considers to not be appropriate to complete participation in the study.
* Ongoing skin issues - Grade I or higher on EPUAP on areas that will be in contact with exoskeleton (European Pressure Ulcer Advisory Panel, 2019)
* Height, width, weight or other anatomical constraints (such as leg length differences) incompatible with the device
* Range of motion (ROM) restrictions in lower extremities, that are incompatible with the device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Time and Level of Assistance (LoA) to don/doff the device [Usability/Feasibility] | Up to 11 weeks
  Level of Assistance (LoA) and time taken to don/doff the device will be measured in every session. LoA will be measured using a 6-item scale, from Total assistance to Independence. Different assistance levels are defined taking into account the degree of participation of the patient and the therapist in performing the activity.
LoA to complete skills for home and community environments [Usability/Feasibility] | Up to 11 weeks
  The participant will attempt a set of skills for home and community environments every session to assess the device's usability. The therapist will record the LoA required to complete each task during every session. The best LoA-Score of all 15 tasks within 3 consecutive training sessions will be recorded and analysed (sessions 2-4, sessions 5-7, sessions 8-10, sessions 11-14, sessions 15-17, sessions 18-20).
Tme to complete Home-Skills-Test and LoA for each task and ti [Usability/Feasibility] | Up to 11 weeks
  A Home-skills-test will be performed by all participants and will consist of 10 of the skills for home and community environments, set out in a sequence to simulate daily life situations. The test will be attempted twice with a 5 min break in between, the best result will be documented. To assure safety, participants will attempt the test with assistance from the therapist as required.
  For all skills of the Home-skills-test, the LoA to complete each task and the time to complete the test will be documented.
Number of steps taken with the device [Usability/Feasibility] | Up to 11 weeks
  The ABLE Exoskeleton device will record the number of steps, walking time, standing time, and walking distance every session. This information will allow insight into the proportion of time spent training per session.
Distance walked with the device [Usability/Feasibility] | Up to 11 weeks
  The ABLE Exoskeleton device will record the number of steps, walking time, standing time, and walking distance every session. This information will allow insight into the proportion of time spent training per session.
Walking time with the device [Usability/Feasibility] | Up to 11 weeks
  The ABLE Exoskeleton device will record the number of steps, walking time, standing time, and walking distance every session. This information will allow insight into the proportion of time spent training per session.
Standing time in the device [Usability/Feasibility] | Up to 11 weeks
  The ABLE Exoskeleton device will record the number of steps, walking time, standing time, and walking distance every session. This information will allow insight into the proportion of time spent training per session.

SECONDARY OUTCOMES:
BORG Scale [Perceived rate of exertion] | Up to 11 weeks
  Measurement of the perceived rate of exertion. The BORG will be tested after the 6 MWT with and without the device. The BORG scale measures the subjective level of intensity in physical work on a 15-grade scale. It ranges from 6 (No exertion at all) to 20 (Maximal exertion).
6-Minute Walk Test (6 MWT) [Gait and function] | Up to 11 weeks
  The 6 Minute Walk Test (6 MWT) measures the distance a person can walk within six minutes. Several conditions are reported to perform the test. For this study we will use a 50 meter track, where the patients are walking back and forth.
10-Meter Walking Test (10 MWT) [Gait and function] | Up to 11 weeks
  The 10 Meter Walk Test (10 MWT) measures the time a person needs to walk 10 meters. The test is performed with a dynamic (flying) start with two-meter acceleration, a timed ten-meter distance and a two-meter deceleration.
Timed up and go test (TUG) [Gait and function] | Up to 11 weeks
  Timed Up and Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around and sit down again. It is a widely used test to assess balance and the risk of falls in different patient groups.
Walking Index for Spinal Cord Injury (WISCI II) [Gait and function] | Up to 11 weeks
  The Walking Index for Spinal Cord Injury (WISCI II) assesses the extent and nature of assistance for walking 10 meters in persons with SCI. Assistance is specified as different combinations of braces, walking aids and physical assistance. The WISCI II consists of 20 levels from inability to walk to the ability to walk 10 meters without any assistance
Spinal Cord Independence Measure (SCIM III) [Gait and function] | Up to 11 weeks
  The Spinal Cord Independence Measure (SCIM) III scale focuses on the ability to perform activities of daily living in persons with SCI. The SCIM III consists of three subscales: Self-Care, Respiratory and Sphincter Management, Mobility (room and toilet) and Mobility (indoors and outdoors, on even surface). A total score of 0 (totally dependent) to 100 (totally independent) points can be achieved
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) [User satisfaction] | Up to 11 weeks
  Used to measure user satisfaction from participants and therapists. The Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) is designed to measure the level of satisfaction and the value people attribute to assistive technologies. It does so using 12 variables which are scored on a 5 point scale in terms of perceived importance and satisfaction. While items 1-8 rate the satisfaction with the device, items 9-12 are for assessing the satisfaction with the service. If the users are not very satisfied with a feature, they are asked to provide specific feedback. The final score is the mean sum scores of all valid responses with a range of 1 (not satisfied at all) to 5 (very satisfied).
Psychosocial Impact of Assistive Devices Scales (PIADS) [Psychosocial impact on participants] | Up to 11 weeks
  The Psychosocial Impact of Assistive Devices Scales (PIADS) is a 26-item (7-point Likert-Scale), self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. It is divided into three subscales: Competence, adaptability and self-esteem. For each of the subscales, typically means are calculated that range from -3 (maximum negative impact) to +3 (maximum positive impact). To have only positive sum scores, the range of the individual scores are shifted to 1 to 7, meaning that sum scores range from 1 *26 (26, maximum negative impact) to 7 *26 (182, maximum positive impact). The PIADS is a responsive measure and sensitive to important variables such as the user's clinical condition, device stigma, and functional features of the device. It has been shown to accurately reflect the self-described experiences of people who use assistive devices
WHO Quality of Life brief form (WHOQOL-BREF) [Participants Quality of Life assessment] | Up to 11 weeks
  The WHO Quality of Life-BREF (WHOQOL-BREF) is the short version of the WHOQOL-100 and is recommended for use when time is restricted or in use in clinical trials. It is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health, psychological health, social relationships and environment. Items are rated on a 5-point Likert scale (low score of 1, high score of 5) to determine a raw item score. Subsequently, the main score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score, with a higher score indicating a higher QOL. When transformed by multiplying by 4, each domain score is then comparable to the scores in the original WHOQOL-100. Self-administration is recommended if the respondent has sufficient ability.
Self-report questionnaire on the perceived impact on general health. | Up to 11 weeks
  Participants' perceptions of the impact on their general health will be evaluated by the completion of a self-report questionnaire on the perceived impact on general health. This questionnaire has been designed by the researchers and intends to identify to what extent participants feel that the ABLE Exoskeleton is ready for home-use.

CONTACTS AND LOCATIONS:
Locations (2):
- Spinal Cord Injury Center | Heidelberg University Hospital, Heidelberg, Germany
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadorf F, Wright MA, Lopez-Matas H, Porras E, Carnicero-Carmona A, Hensel C, Franz S, Weidner N, Vidal J, Opisso E, Rupp R. User-centered design of a personal-use exoskeleton: a clinical investigation on the feasibility and usability of the ABLE Exoskeleton device for individuals with spinal cord injury to perform skills for home and community environments. Front Neurosci. 2024 Sep 26;18:1437358. doi: 10.3389/fnins.2024.1437358. eCollection 2024. PMID 39391753